CLINICAL TRIAL: NCT02990702
Title: Retroclavicular Approach vs Infraclavicular Approach for Brachial Plexus Block in Obese
Brief Title: Retroclavicular Approach vs Infraclavicular Approach for Brachial Plexus Block in Obese Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Bora Bilal, Assistant Proffesor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 31
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Forearm Injuries; Hand Injuries
Keywords: Infraclavicular block; Retroclavicular block; Ultrasound
MeSH Terms: conditions — Forearm Injuries; Hand Injuries | interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided retroclavicular block (Active Comparator): Ultrasound guided retroclavicular block group patients (Group R) will receive 30 cc %0.5 Bupivacaine
  Interventions: Other: Ultrasound guided retroclavicular block; Other: Ultrasound guided coracoid infraclavicular block; Drug: Bupivacaine; Device: Ultrasound
- Ultrasound guided infraclavicular block (Active Comparator): Ultrasound guided coracoid infraclavicular block group patients (Group C) will receive 30 cc %0.5 Bupivacaine
  Interventions: Other: Ultrasound guided retroclavicular block; Other: Ultrasound guided coracoid infraclavicular block; Drug: Bupivacaine; Device: Ultrasound

INTERVENTIONS:
Other: Ultrasound guided retroclavicular block — Ultrasound guided retroclavicular block for forearm or hand surgery
  Other Names: Group R
Other: Ultrasound guided coracoid infraclavicular block — Ultrasound guided infraclavicular block for forearm or hand surgery
  Other Names: Group C
Drug: Bupivacaine
Device: Ultrasound

SUMMARY:
The retroclavicular approach for brachial plexus anesthesia requires an optimal angle between the needle and the ultrasound beam. Retroclavicular approach has already been proven effective and safe in the past. The general objective is to provide a formal comparison between the retroclavicular approach and coracoid infraclavicular approach for brachial plexus anaesthesia. This study should represent the differences between the two techniques.

DETAILED DESCRIPTION:
Classic infraclavicular approach of the brachial plexus involves a needle puncture below the clavicle and advancing the needle with a 45-60 degree angle from cephalad to caudad. The aim is to advanced the block needle posterior to the axillary artery and to deposit the local anesthetic at that point, near the posterior cord. A "U" shaped spread around the artery should ensure distribution around all three cords. Ultrasound guidance is highly recommended and neurostimulation is optional.

The retroclavicular approach is a variant to this classical technique. Ultrasound probe is positioned initially below the clavicle in a manner similar to the classic approach but is then rotated in a clockwise fashion (right arm) or counter-clockwise fashion (left arm) for about 25-35 degrees. The puncture site is just behind the clavicle at the most lateral point available. If initial entry point is optimal, needle direction is then parallel to ultrasound probe. The final aim and position of block needle is identical to classical approach. Entry point ensures a parallel alignment of the needle and the ultrasound beam, thus enabling almost perfect visualization of both artery, cords and block needle. This is turn optimizes safety, rapidity of technique, efficiency and efficacy.

It is recognized that regional anesthesia is more difficult to perform in obese patients. Anatomic landmarks are harder to localize in this population and ultrasound guidance is more difficult because of the attenuation of the ultrasound beam by adipose tissue. The complication rate of regional techniques is also reported to be higher in the obese patient population.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* BMI>30
* Forearm- Hand surgery

Exclusion Criteria:

* <18 years
* Local infection
* Coagulopaty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Technique duration | Measured directly during the procedure with a chronometer.
  The performance time corresponds to the sum of imaging time and needling time. It is expressed in minutes. Analysis of the primary outcome: performance time will be analyzed with a non-inferiority test of the averages, with the objective of finding that the experimental retroclavicular approach is no longer to perform than the coracoid infraclavicular approach.
Surgery completion under regional block | Success is defined at end of surgery for which block was done, generally within 1 to 3 hours after block is performed
  Success rate is defined as the completion of the intended surgery under regional anaesthesia with retroclavicular block without the need for a rescue technique.

SECONDARY OUTCOMES:
Sensorial block progression | Assessed 10, 20 and 30 minutes after block completion
  Progress of the sensory block in the distribution of the radial, median, ulnar, musculocutaneous, and medial cutaneous nerves of the forearm and hand at 10, 20 and 30 minutes after block completion. The scale used is: 0:no sensitive block, 1:analgesia (loss of pain but not tactile sensation), 2:anesthesia (loss of pain and tactile sensation).
Motor Block Progression | Assessed 10, 20, 30 minutes after the block completion
  Progress of the motor block in the distribution of the radial, median, ulnar, musculocutaneous nerves of the forearm and hand at 10, 20, and 30 minutes after block completion. The scale used is: 0: no motor block, 1: paresis, 2: paralysis. No units are attached to this scale.
Needle visualization | Assessed one week after study completion
  Procedures will be recorded and reviewed simultaneously after study completion by 2 independent anesthesiologists skilled in US-guided regional anesthesia using a 5-point Likert scale to rate needle visibility (1=very poor,2=poor,3=fair,4=good,5=very good)

IPD SHARING:
Plan to Share IPD: No